CLINICAL TRIAL: NCT06903897
Title: Improving Chronic Disease Outcomes Across the Lifespan by Addressing Structural Racism
Brief Title: Social Needs Screening and Chronic Diseases Study (WE CARE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Boston University (Other); Boston Medical Center (Other); Family Health Center of Worcester (Unknown)
Responsible Party: Principal Investigator, Arvin Garg, Professor of Pediatrics, University of Massachusetts, Worcester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00001499; 1R01NR020752-01 (NIH)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hyperlipidemias; Diabetes; Depression; Pediatric Asthma; Hypertension
Keywords: Basic Needs; Social Determinants of Health; Screening tools; Antiracism
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus; Depression; Hypertension

STUDY DESIGN:
Intervention Model Description: A stepped wedge cluster Randomized Controlled Trial (RCT) will be conducted whereby the investigators will provide the intervention to all participants but stagger the timing of introduction to compare practices to one another and to compare practices to themselves, before and after implementation of the WE CARE model. This design minimizes the risk of contamination at the practice level, equitably implements the model in all clinical sites (vs. withholding in a traditional RCT design) and allows the investigators to simultaneously test the implementation and effectiveness of WE CARE in all study sites. Research staff at the study sites will abstract medical records (of adults and children with chronic diseases that are eligible (have diagnosis of hypertension, diabetes mellitus, hyperlipidemia, or depression for adults or have diagnosis of asthma for children) for administration of the WE CARE screener on a regular basis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care - Control (Active Comparator): Participants in the usual care group receive standard pediatric care. In this study, participants in the Usual Care arm are a historical cohort of patients who meet eligibility criteria and are identified retrospectively from the Electronic Health Records. As such the investigators have registered this study on Clinical Trial.gov prior to the implementation of the active WE CARE experimental arm.
  Interventions: Other: Standard Pediatric Care
- WE CARE Implementation Arm (Experimental): The study team will work with clinic staff and leadership to implement the WE CARE protocol at each clinical site.
  Interventions: Other: WE CARE SDOH System

INTERVENTIONS:
Other: WE CARE SDOH System — The WE CARE System: A family-centered, highly efficacious approach for addressing adverse SDOH in the clinical setting. Arvin Garg, MD, MPH developed and conceptualized the WE CARE (Well-Child care visit, Evaluation, Community Resources, Advocacy, Referral, Education) intervention in 2005. This approach relies on existing clinical processes and infrastructure and social service resources, thereby making implementation, dissemination, and sustainability feasible. The intervention components include brief training of the clinical team; administration of a short screening tool to parents/patients identifying their desire for help with specific unmet social needs; and provider/clinic staff access to a physical or electronic family resource book containing community- resource listings. Providers generate referrals for families who indicate that they want help with unmet social needs on the WE CARE screener. Existing staff members may assist patients in connecting to referred resources.
  Arms: WE CARE Implementation Arm
Other: Standard Pediatric Care — Standard pediatric care includes any existing screening practices, which can vary at each clinic.
  Arms: Usual Care - Control

SUMMARY:
The goal of this clinical trial is to learn if the implementation of the WE CARE social determinants of health (SDOH) screening and referral intervention with an antiracist lens in primary care settings can lead to a meaningful decrease in chronic disease by monitoring conditions such as hypertension, diabetes, depression, hyperlipidemia, and asthma through clinical measures. The main question it aims to answer is:

Does the WE CARE SDOH screening and referral intervention applying an antiracism lens informed implementation strategies have the potential to reduce racial/ethnic health inequities in chronic diseases for minoritized patients?

DETAILED DESCRIPTION:
With a multidisciplinary team of social determinants of health (SDOH), implementation, antiracism, community-engaged, and practice-based researchers, the investigators will apply an antiracism framework to an existing evidence-based SDOH screening and referral system and develop a holistic implementation toolkit aimed at reducing bias and mitigating unequal treatment for families of color. The investigators will first conduct qualitative interviews with adult patients and caregivers to understand their experiences with racism and discrimination within the context of their experiences with screening and referral for SDOH; the investigators will then share their findings with stakeholders (e.g., clinic directors, community agency leaders, health system leaders, Medicaid leaders) and elicit their ideas on how best to address these issues within the systems they lead. Subsequently, the investigators will refine the WE CARE implementation protocol using this stakeholder input with the guidance of antiracism and implementation experts. The investigators will then implement the refined WE CARE protocol in family medicine clinics since adverse SDOH impact the whole family unit; it will also allow them to examine WE CARE's impact on improving health outcomes for racialized groups across the life course. The investigators will conduct a hybrid effectiveness-implementation study with a stepped wedge cluster RCT design in three large family medicine clinics (including 2 health centers) that serve racially/ethnically diverse low-income families from Worcester, Massachusetts. The specific aims are to:

* Aim 1: Refine the WE CARE implementation protocol using an antiracism lens and community engagement approach to: (a) conduct key informant interviews with families to identify racism and discrimination related barriers to SDOH screening/referral; (b) present these barriers to systems-level stakeholders to elicit input on strategies to address patient concerns; and 3) create an antiracist informed toolkit for the implementation of SDOH screening/referral.).*
* Aim 2: Deploy the refined WE CARE protocol in family medicine practices and assess implementation outcomes including equity, appropriateness, and patient-centeredness
* Aim 3: Conduct a clinical trial to evaluate the effectiveness of the refined WE CARE protocol on prevalent pediatric and adult chronic diseases (e.g., asthma, diabetes, hyperlipidemia, hypertension, depression) outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adults and children with diagnosed chronic diseases (hypertension, diabetes mellitus, hyperlipidemia, asthma, or depression) who receive Family Medicine care at one of the study sites.
* Children (<18 years of age) with a diagnosis of asthma.
* Adult patients (18 years or older) with a diagnosis of diabetes mellitus, hypertension, hyperlipidemia and/or depression.

Exclusion Criteria:

* In adults (>18 years of age), those without one or more of the following diagnoses as recorded by ICD-10 codes in their EHR: hypertension, hyperlipidemia, diabetes mellitus, or depression.
* In children (<18 years of age), those without a diagnosis of asthma.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68000 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (BP) measurements | Every 3 months for up to 3 years
  Systolic and diastolic blood pressure measurements collected at all routine and follow-up visits for adults.

SECONDARY OUTCOMES:
LDL-C measurements | Every 3 months for up to 3 years
  Laboratory assessment for lipid (LDL-C) levels for adult patients with hyperlipidemia.
HbA1c measurements | Every 3 months for up to 3 years
  Laboratory assessment for Hba1C levels for diabetes patients.
Emergency department visits | Every 3 months for up to 3 years
  All ED visits whether or not they lead to a hospitalization for children and adults. (total, Asthma related, non-emergent)
Hospitalizations | Every 3 months for up to 3 years
  Hospitalizations for children and adults (total, ACSC, Asthma related, CVD)

OTHER OUTCOMES:
Body mass index | Every 3 months for up to 3 years
  Clinical BMI assessment
Clinic visit adherence | Every 3 months for up to 3 years
  Clinic visit attendance (appointment-keeping/no-shows)
Adverse social determinants of health (SDOH) | Every 3 months for up to 3 years
  Number/types of patient's unmet social needs
Social determinants of health (SDOH) screening | Every 3 months for up to 3 years
  Number of screeners given by providers to patients.
Provider referrals | Every 3 months for up to 3 years
  Number/types of referrals to social services given by providers to patients.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - (Benedict) UMass Memorial Medical Center - Adult Primary Care, Worcester, Massachusetts
  - UMass Memorial Medical Center - Hahnemann Campus, Worcester, Massachusetts
  - Family Health Center of Worcester, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No